CLINICAL TRIAL: NCT06534814
Title: Hebei Medical University
Brief Title: Development and Application of an Artificial Intelligence-driven Accurate Identification Model for Gastric Cancer Lymph Node Metastasis
Status: Recruiting | Type: Observational
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Qun Zhao, Professor, Hebei Medical University
Other Study IDs: FUTURE08
Record Dates: First submitted 2024-07-25; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: The Primary Focus of This Study is on Gastric Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: AI-Driven Identification Model for Gastric Cancer Lymph Node Metastasis (AID-GLNM) — The AI-Driven Identification Model for Gastric Cancer Lymph Node Metastasis (AID-GLNM) intervention involves the development and application of an advanced artificial intelligence (AI) system specifically designed to enhance the identification and characterization of lymph node metastasis in patients diagnosed with gastric cancer.

SUMMARY:
The clinical trial titled "Development and Application of an Artificial Intelligence-Driven Accurate Identification Model for Gastric Cancer Lymph Node Metastasis" aims to enhance the detection and treatment of gastric cancer through the utilization of cutting-edge artificial intelligence (AI) technology. This study will develop an AI-driven model designed to accurately identify lymph node metastasis in patients with gastric cancer, which is crucial for staging the disease and planning effective treatment strategies.

The trial will involve a multidisciplinary team of oncologists, radiologists, data scientists, and AI experts who will collaborate to create a robust and precise identification system. Participants will undergo standard diagnostic procedures, and the AI model will analyze imaging and pathological data to predict lymph node involvement.

By comparing the AI model's predictions with traditional diagnostic methods, the study seeks to validate the model's accuracy and efficiency. This approach is expected to improve early detection rates, reduce diagnostic errors, and ultimately lead to better clinical outcomes for patients with gastric cancer. The successful implementation of this AI-driven model could revolutionize the current standards of care and serve as a blueprint for integrating AI technologies in other cancer diagnoses and treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Gastric Cancer: Confirmed diagnosis of gastric cancer, either newly diagnosed or recurrent.
2. Lymph Node Involvement: Suspected or confirmed involvement of lymph nodes, as indicated by imaging studies or pathology reports.
3. Age: Patients aged 18 years or older.
4. Performance Status: An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2, indicating a functional status that allows participation in the study.
5. Informed Consent: Ability to provide written informed consent to participate in the study.

Exclusion Criteria:

1. Pregnancy or Lactation: Pregnant or lactating women, due to potential risks to the fetus or infant.
2. Severe Comorbid Conditions: Presence of severe comorbid medical conditions that could interfere with the study or pose additional risks.
3. Previous AI-Driven Diagnostic Intervention: Prior use of any AI-driven diagnostic models specifically for gastric cancer lymph node metastasis.
4. Inability to Comply: Inability or unwillingness to comply with study procedures, including follow-up visits and data collection.
5. Mental or Cognitive Impairment: Conditions that impair the ability to provide informed consent or participate effectively in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population for the clinical trial titled "Development and Application of an Artificial Intelligence-Driven Accurate Identification Model for Gastric Cancer Lymph Node Metastasis (AID-GLNM)" will consist of patients diagnosed with gastric cancer, with a focus on those exhibiting lymph node involvement.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
Identification of metastatic lymph nodes | 2025-12-31
  A prediction model based on artificial intelligence technology was constructed to accurately identify metastatic perigastric lymph nodes before surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery, Shijiazhuang, Hebei, China